CLINICAL TRIAL: NCT02178150
Title: Effect of Magnesium Supplementation on Metabolic Profile and Sex Hormone Levels in Overweight Women With Polycystic Ovary Syndrome.
Brief Title: Effect of Magnesium Supplementation on Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Associate Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18201
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Magnesium; Insulin Resistance; Lipid profile; Sex hormones; Inflammatory factors
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Oxide (Active Comparator): magnesium tablets, 250 milligram magnesium, 8 weeks, every day 1 tablet
  Interventions: Dietary Supplement: Magnesium Oxide
- Placebo (Placebo Comparator): Placebo tablets, the same in color, odor and appearance with magnesium tablets, 8 weeks, one tablet every day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium Oxide — This is a double-blind randomized clinical trial which will be started at June 2014 and end on June 2015 in Isfahan city. Serum insulin level is considered as a key variable and the sample size was calculated to be 70 persons (35 persons for control group and 35 persons for patient group). Patient group will receive magnesium supplement (250 milligram) and the other group will receive placebo which is similar to the magnesium tablets in color, odor and appearance both for 8 weeks. All subjects will complete 4 physical activity and 4 dietary records. Outcome measurements including metabolic and inflammatory profiles,sex hormone levels will be measured at the beginning and end of the study as well as anthropometric measurements.
  Arms: Magnesium Oxide
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind randomized clinical trial which will start at June 2014 and end on June 2015 in Isfahan city. Serum insulin level is considered as a key variable and the sample size calculated 70 persons (35 persons for control group and 35 persons for patient group). Patient group will receive magnesium supplement (250 milligram) and the other group will receive placebo which is similar to the magnesium tablets in color, odor and appearance both for 8 weeks. All subjects will complete 4 physical activity and 4 dietary records. Outcome measurements including sex hormone levels, metabolic and inflammatory profiles will be measured at the beginning and end of the study as well as anthropetric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Having PCOS according to the Rotterdam criteria,
* Age between 20-45 years,
* Lack of pregnancy and lactation,
* Not having certain regime during last 3 months,
* Non-smoking,
* Not having diseases, including: diabetes, cardiovascular , hepatic, renal and thyroid,
* Not taking supplements,
* Being overweight (Kg / m 25 ≤ BMI)

Exclusion Criteria:

* Hormone Therapy,
* Pregnancy and lactation during the study,
* Severe weight loss (more than 2.5 kg per month) during the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serum insulin level | 8 Weeks

SECONDARY OUTCOMES:
Insulin Resistance | 8 weeks
Fasting Blood Sugar | 8 weeks
Quantitative insulin sensitivity check index (Quicki) | 8 weeks
HOMA-IR | 8 weeks
HOMA-B | 8 weeks
High Density Lipoprotein | 8 weeks
Low Density Lipoprotein | 8 weeks
Triglyceride | 8 weeks
Total Cholesterol | 8 weeks
Androgen | 8 weeks
Testosterone | 8 weeks
C-Reactive Protein | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Esmaeilzadeh, professor, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Farsinejad-Marj M, Azadbakht L, Mardanian F, Saneei P, Esmaillzadeh A. Clinical and Metabolic Responses to Magnesium Supplementation in Women with Polycystic Ovary Syndrome. Biol Trace Elem Res. 2020 Aug;196(2):349-358. doi: 10.1007/s12011-019-01923-z. Epub 2020 Jan 20. PMID 31960275